CLINICAL TRIAL: NCT02148003
Title: Effect of the Temperature Used in Thermal Radiofrequency Ablation on Outcomes of Lumbar Facets Medial Branches Denervation Procedures: A Randomized Double-Blinded Trial
Brief Title: Effect of the Temperature Used in Thermal Radiofrequency Ablation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated by Principal Investigator
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-1470
Record Dates: First submitted 2014-04-22; First posted 2014-05-28 (Estimated); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RFA at 90 degrees Celsius (Active Comparator): Radiofrequency ablation (RFA) of the lumbar facets nerve supply will be performed at 90 degrees Celsius
  Interventions: Procedure: RFA at 90 degrees Celsius; Device: C-arm guided 20-gauge radiofrequency needle
- RFA at 80 degrees Celsius (Active Comparator): Radiofrequency ablation (RFA) of the lumbar facets nerve supply will be performed at 80 degrees Celsius
  Interventions: Procedure: RFA at 80 degrees Celsius; Device: C-arm guided 20-gauge radiofrequency needle

INTERVENTIONS:
Procedure: RFA at 90 degrees Celsius — Ablation at 90 degrees Celsius is defined as radiofrequency ablation of the lumbar facets nerve supply will be performed at 90 degrees Celsius
  Arms: RFA at 90 degrees Celsius
Procedure: RFA at 80 degrees Celsius — Ablation at 80 degrees Celsius is defined as radiofrequency ablation of the lumbar facets nerve supply will be performed at 80 degrees Celsius
  Arms: RFA at 80 degrees Celsius
Device: C-arm guided 20-gauge radiofrequency needle — Needles will be adjusted to optimize sensory and motor stimulation.

SUMMARY:
This study will determine if lumbar facets medial branches RFA at 90 degrees Celsius provides more overall pain relief (i.e., percent of improvement), when compared to ablation at 80 degrees Celsius with no additional adverse events.

DETAILED DESCRIPTION:
Chronic lower back pain (CLBP) is a significant health care issue in the United States and the world. CLBP contributes to decreased quality of life, decreased function and increased utilization of health care resources. The causes of CLBP tend to be multi-factorial. Arthropathy of the lumbar facet joints is thought to be a common etiology (15-45%). Radiofrequency Ablation (RFA) of the medial branch nerve of the facet joint is a well-established treatment modality used to decrease facet joint pains. However, a wide range of temperature is being used (70-90 degrees Celsius). In addition, the optimal temperature that provides the best patient outcomes with the least side effects is not well established in the pain management literature.

This study will determine if lumbar facets medial branches RFA at 90 degrees Celsius provides more overall pain relief (i.e., percent of improvement), when compared to ablation at 80 degrees Celsius with no additional adverse events. Furthermore, ablation of the lumbar facets nerve supply at 90 degrees Celsius will provide better improvement in the functionality level, general mood and quality of life as measured by VAS ( Visual Analog Scale) pain score, Pain Disability Index (PDI), McGill Pain questioner scores and Beck Inventory (BI) scores as those receiving the ablation at 80 degrees Celsius. Also, it is associated with less opioid consumption, no additional unwanted adverse events and/or complications along with less need to repeat RFA procedure over one year period.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years-old
* Subjects who are able to give informed consent and to understand and comply with study requirements.
* Predominantly axial low back pain ≥ 3 months in duration with no radicular pain below the knee that failed to conservative therapy.
* Subjects who have chronic back pain attributed to lumbar facet joints arthropathy based on clinical evaluation (paraspinal tenderness and/or facet loading test in the absence of signs and symptoms suggestive of focal neurological deficits).
* No history of previous back surgery at the intended treatment levels.
* Adequate response to the diagnostic blocks without the use of steroids at the same levels of the intended block (Defined as ≥ 75% pain relief).
* Patients who will undergo RFA of 3-4 lumbar facet medial branches on one side only.

Exclusion Criteria:

* Subjects who decline to provide written consent or follow-up.
* Subjects who have a history of adverse reactions to local anesthetic.
* Subjects who are pregnant.
* Subjects with bleeding disorders or active anticoagulation that cannot be stopped for few days close to the time of the procedure.
* Subjects who have an active systemic or local infection.
* Presence of radicular pain below the knee.
* Patients who have other specific etiology of low back pain (e.g. significant spinal canal stenosis or grade 2 or 3 spondylolisthesis).
* Secondary gain (i.e., ongoing litigation, worker's compensation or other financial incentives)
* Psychopathology including depression, somatization or poor coping skills
* Physical factors including non-sedentary lifestyle, e.g.; morbid obesity (BMI > 35kg/m2).
* History of previous RFA at the same level(s) in the previous 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagy Mekhail, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RFA at 90 Degrees Celsius | RFA at 80 Degrees Celsius
Started | 60 | 60
Completed | 59 | 58
Not Completed | 1 | 2
Not completed — Failed inclusion criteria | 1 | 0
Not completed — Met exclusion criteria | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 58 patients received RFA at 80°C and 59 patients received RFA at 90°C.
Groups:
- Total: Total of all reporting groups
Arm/Group | RFA at 90 Degrees Celsius | RFA at 80 Degrees Celsius | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Continuous [Mean (Standard Deviation); unit: year] | 57 (13) | 61 (14) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race data was not collected.. Population: Race data was not collected..
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28 (4) | 28 (4) | 28 (4)
Smoking history [Count of Participants; unit: Participants] — Any use of tobacco before the procedure
  Participants
    Yes | 19 | 15 | 34
    No | 40 | 43 | 83
Diabetes history [Count of Participants; unit: Participants] — Any medical history of type II diabetes before the procedure
  Participants
    Yes | 6 | 12 | 18
    No | 53 | 46 | 99

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Score 30-day After Procedure
Description: The primary outcome was the Visual Analog Scale (VAS) pain score at 30-day follow-up visit, which was collected by patients marking a position on a strip to indicate the intensity of their pain. The locations patients marked are translated into a score from 0-100, with 0 being no pain and 100 corresponding to the worst imaginable pain.
Time Frame: 30 days after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RFA at 90 Degrees Celsius | RFA at 80 Degrees Celsius
Number analyzed (Participants) | 59 | 58
units on a scale | 50.4 (31.4) | 47.2 (30.5)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the end of procedure to the 1-year follow-up.
Arm/Group | RFA at 90 Degrees Celsius | RFA at 80 Degrees Celsius
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58
Other Adverse Events (participants affected / at risk) | 0/59 | 0/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RFA at 90 Degrees Celsius (N=59) | RFA at 80 Degrees Celsius (N=58)
Persistent Parethesia (Surgical and medical procedures) | 0 | 0
Nerve injuries (Surgical and medical procedures) | 0 | 0
Bleeding (Surgical and medical procedures) | 0 | 0
Infection (Surgical and medical procedures) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT02148003/Prot_SAP_000.pdf